CLINICAL TRIAL: NCT06809855
Title: The Effectiveness of Using a Single Post-operative Intramuscular Dexamethasone Injection on Patients with Surgical Extraction of Lower Third Molar(Split Mouth Technique)
Brief Title: The Effectiveness of Using a Single Post-operative Intramuscular Dexamethasone Injection on Patients with Surgical Extraction of Lower Third Molar
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yassir R. Al-khannaq (Other)
Responsible Party: Sponsor-Investigator, Yassir R. Al-khannaq, lecturer Dr., University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 997124
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Dexamethasone Administration; Post Extraction Complication
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Each patient resembles the study group in which the patient is injected intramuscularly by a single dose 8mg dexamethasone immediate postoperatively after removal of impacted mandibular third molar on one side and control group on which the impacted mandibular third molar on the other side is removed without usage of 8mg dexamethasone.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- dexamethasone immediate injection postoperatively (Active Comparator): intramuscular injection of a single dose 8mg dexamethasone immediate postoperatively after removal of impacted mandibular third molar
  Interventions: Drug: Dexamethasone
- no intervention (No Intervention)

INTERVENTIONS:
Drug: Dexamethasone — single 8mg post-operative intramuscular injection
  Arms: dexamethasone immediate injection postoperatively

SUMMARY:
Evaluating the effectiveness of using a single immediate postoperative intramuscular Dexamethasone injection on pain, swelling, trismus and tissue healing in the first seven days.

Methods: A split mouth technique on 16 patients with bilateral similar impacted mandibular third molar were extracted; one side was given 8mg intramuscular injection of dexamethasone (study group) and the other side wasn't given injection (control group) and compare of the two sides were done in the following seven days.

ELIGIBILITY:
Inclusion Criteria:

* bilateral similar impacted lower third molar
* willing to do surgical extraction

Exclusion Criteria:

* Patients who are not fulfill the inclusion criteria
* allergic to dexamethasone
* who has medical diseases
* taking any medications
* pregnant or lactating women

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-16 (Actual)

PRIMARY OUTCOMES:
post operative pain changes | each participant was seen at 1st, 3rd and 7th post-operative days
  measurement of change in pain on visual scale analog from 10 to 1 , 10 mean the worst pain and 1 is least pain
Change in post operative swelling | each participant was seen at 1st, 3rd and 7th post-operative days
  The swelling was measured between two points marked on skin in millimeters using ruler
Post operative Change in mouth opening | each participant was seen at 1st, 3rd and 7th post-operative days
  The distance between upper and lower incisors was measured in millimeters using ruler

SECONDARY OUTCOMES:
Tissue healing | Healing was assessed on the 7th postoperative day
  Healing of extraction site was assessed by using Landry, Turnbull and Howley index

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral and Maxillofacial Surgery, College of Dentistry, University of Baghdad, Baghdad, Iraq